CLINICAL TRIAL: NCT02777086
Title: Sustainable HIV Risk Reduction Strategies for Criminal Justice (CJ) Systems
Brief Title: Sustainable HIV Risk Reduction Strategies for Probationers
Acronym: DRR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DA25885-1506-060-1508
Record Dates: First submitted 2016-04-20; First posted 2016-05-19 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Health Behavior
Keywords: HIV; Risk Behaviors; Decision-making
MeSH Terms: conditions — Health Behavior; Risk-Taking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- StaySafe (Experimental): Participants are asked to complete 12 brief, self-administered tablet computer sessions designed to improve decision-making around health risk behaviors. Sessions typically take about 10 minutes each to complete and are scheduled prior to or after probationer group or individual appointments at their probation facility. Sessions are scheduled about once per week.
  Interventions: Behavioral: StaySafe
- Comparison (No Intervention): Participants are asked to complete baseline, 3-month and 6-month surveys but are not asked to complete StaySafe sessions or other alternate activities.

INTERVENTIONS:
Behavioral: StaySafe — StaySafe is a self-administered tablet computer app designed to improve decision-making around health risk behaviors.
  Arms: StaySafe

SUMMARY:
The purpose of the Texas Christian University (TCU) Disease Risk Reduction (DRR2) Project is to develop and test a self-administered tablet computer app, StaySafe, for probationers under community supervision that is designed to improve decision-making skills around health risk behaviors, especially involving HIV and hepatitis B & C risks. StaySafe utilizes materials and concepts adapted from an earlier, group-based curriculum, WaySafe, designed to increase positive decision-making skills for offenders in the last phase of their prison-based substance abuse treatment before transitioning back to the community.

DETAILED DESCRIPTION:
The purpose of the TCU DRR2 project is to adapt ideas and concepts from an in-prison, group-based curriculum designed to improved decision-making skills around health risk behaviors for incarcerated offenders in the last phase of substance abuse treatment for a self-administered computer app that targets probationers under community supervision. Programming for HIV in probation settings is limited and this project aims to address needs with an easy to use computer app that is designed to improve decision-making about health risks among probationers in the community. The computer app utilizes an evidence-based schema called WORKIT and is based on a dual processing model of judgment and decision-making that includes vicarious and virtual learning approaches and repetition in order to learn and practice the schema and move it from slower analytical processing to faster experiential processing.

StaySafe includes 12 brief sessions, each of which takes about 10 minutes to complete. Nine of the sessions utilize the WORKIT model and three session use a participant choice activity in which probationers can choose from among several informational activities designed to reinforce lessons learned and provide some variation to completing WORKIT sessions. The first session includes an introduction to using the app on the tablet and guides the participant through a WORKIT session. In each subsequent WORKIT session, the participant chooses a relevant problem to work on during that session from a list of problems. A brief video is then shown in which two people are having a conversation around the problem and make a decision. The participant rates the decision before working through the WORKIT process around the chosen problem. This involves determining what the problem is, who is affected by the problem and who can help with the problem, then identifying options to address the problem, rating the options, knowing what option to choose, imagining the steps to carry out the option, and then testing the results. Sessions are typically scheduled about every two weeks.

Participants are recruited by research staff for the study from probation offices where substance abuse groups are conducted. All assessment and StaySafe sessions are administered by research staff at the probation facility when probationers otherwise report for meetings or groups. Compensation for time involved in the study is provided in terms of payments toward probation fees. After an Institutional Review Board (IRB)-approved consent procedure, participants are scheduled for a baseline survey that takes about 30 minutes to complete. After the baseline survey is completed, participants are randomly assigned to either the StaySafe condition or a comparison condition. Participants in the StaySafe condition are then scheduled for their first StaySafe session typically within a week and are asked to complete twelve sessions within the next 6 months, followed by 6-month and 12-month follow-up surveys. Participants randomly assigned to a comparison condition are informed that they will be contacted in about 6 months to schedule a 6-month survey and again for a 12-month survey.

ELIGIBILITY:
Inclusion Criteria:

* On probation
* Has received prior drug treatment from an in-prison, residential, or intensive outpatient program
* Can read at the 4th grade level

Exclusion Criteria:

* Does not have 6 months of probation left
* Is not a sex offender
* Does not have a serious mental health diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne E Lehman, PhD, Principal Investigator — Institute of Behavioral Research, Texas Christian University
Locations (3):
- United States (3):
  - Dallas County CSCD, Dallas, Texas
  - Tarrant County CSCD, Fort Worth, Texas
  - Harris County CSCD, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data files will be prepared at the conclusion of the study to be embargoed for two years after the end of grant funding for archiving in the National Addiction and HIV Data Archives (NAHDAP) funded by the National Institute on Drug Abuse (NIDA) and hosted by the Inter-university Consortium for Political and Social Research, which is part of the University of Michigan's Institute for Social Research. NAHDAP archives and preserves data produced by research grants to support secondary data analysis by other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: two years after conclusion of the study
Access Criteria: no restrictions

REFERENCES:
- [Derived] Joe GW, Lehman WEK, Yang Y, Knight K. The Effectiveness of the StaySafe Intervention Using a Paradigm for Predicting Missing Outcome Data. Eval Health Prof. 2025 Sep;48(3):374-383. doi: 10.1177/01632787231212462. Epub 2023 Nov 13. PMID 37956984
- [Derived] Joe GW, Lehman WEK, Pankow J, Wiese A, Knight K. Decision-Making Styles as a Moderator on the Efficacy of the StaySafe Tablet Intervention. Subst Use Misuse. 2023;58(9):1132-1142. doi: 10.1080/10826084.2023.2212301. Epub 2023 May 15. PMID 37184071

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruiting for the study began in September, 2015 and extended through February, 2019. Recruitment occurred in probation offices in two large counties in Texas and two residential substance abuse treatment centers for people on probation.
Period: Overall Study
Arm/Group | StaySafe | Comparison
Started | 261 | 250
Completed | 165 | 151
Not Completed | 96 | 99
Not completed — Lost to Follow-up | 96 | 99

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | StaySafe | Comparison | Total
Number analyzed (Participants) | 261 | 250 | 511
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 261 | 250 | 511
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 113 | 249
  Male | 125 | 137 | 262
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 80 | 80 | 160
  Not Hispanic or Latino | 179 | 170 | 349
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 87 | 77 | 164
  White | 138 | 153 | 291
  More than one race | 29 | 14 | 43
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 261 | 250 | 511
HIV Knowledge Confidence [Mean (Standard Deviation); unit: units on a scale] — Questionnaire measure of knowledge, confidence & motivation around HIV knowledge. Values range from 10 to 50 with higher scores indicating higher knowledge, confidence & motivation.
  units on a scale | 40.2 (7.2) | 40.0 (7.4) | 40.1 (7.3)
Avoiding risky sex [Mean (Standard Deviation); unit: units on a scale] — Questionnaire measure of knowledge, confidence, and motivation in avoiding risky sex behaviors. Values range from 10 to 50 with higher scores indicating higher knowledge, confidence & motivation.
  units on a scale | 41.1 (7.3) | 40.6 (7.4) | 40.8 (7.3)
HIV Services & Testing [Mean (Standard Deviation); unit: units on a scale] — Questionnaire measure of knowledge, and motivation around getting tested for HIV and obtaining HIV services. Values range from 10 to 50 with higher scores indicating higher knowledge, confidence & motivation.
  units on a scale | 41.7 (6.4) | 41.8 (6.5) | 41.8 (6.5)
Risk Reduction Skills [Mean (Standard Deviation); unit: units on a scale] — Questionnaire measure of knowledge, confidence and motivation around risk reduction skills. Values range from 10 to 50 with higher scores indicating higher knowledge, confidence & motivation.
  units on a scale | 42.7 (5.8) | 42.4 (6.0) | 42.5 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: HIV Knowledge Confidence
Description: Questionnaire measure of knowledge, confidence & motivation around HIV knowledge. Values range from 10 to 50 with higher scores indicating higher knowledge, confidence & motivation.
Time Frame: 3-months
Population: Outcome analyses were computed on participants in the StaySafe and Comparison groups who had a baseline and a 3-month follow-up survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | StaySafe | Comparison
Number analyzed (Participants) | 165 | 151
units on a scale | 42.9 (5.4) | 40.5 (7.1)
Statistical Analysis 1: Comparison: StaySafe vs Comparison; 3-month outcome measures were compared between the StaySafe and Comparison groups controlling for the baseline measure using generalized linear models; Test type: Superiority; p < .001, ANCOVA

2. Primary Outcome: Avoiding Risky Sex
Description: Questionnaire measure of knowledge, confidence, and motivation in avoiding risky sex behaviors. Values range from 10 to 50 with higher scores indicating higher knowledge, confidence & motivation.
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | StaySafe | Comparison
Number analyzed (Participants) | 165 | 151
units on a scale | 43.1 (5.6) | 41.3 (7.1)

3. Primary Outcome: HIV Services & Testing
Description: Questionnaire measure of knowledge, and motivation around getting tested for HIV and obtaining HIV services. Values range from 10 to 50 with higher scores indicating higher knowledge, confidence & motivation.
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | StaySafe | Comparison
Number analyzed (Participants) | 165 | 151
units on a scale | 44.3 (5.3) | 42.1 (5.9)

4. Primary Outcome: Risk Reduction Skills
Description: Questionnaire measure of knowledge, confidence and motivation around risk reduction skills. Values range from 10 to 50 with higher scores indicating higher knowledge, confidence & motivation.
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | StaySafe | Comparison
Number analyzed (Participants) | 165 | 151
units on a scale | 44.3 (4.7) | 43.0 (5.6)

ADVERSE EVENTS:
Time Frame: 6 months
Description: No adverse events were observed
Arm/Group | StaySafe | Comparison
All-Cause Mortality (participants affected / at risk) | 0/261 | 0/250
Serious Adverse Events (participants affected / at risk) | 0/261 | 0/250
Other Adverse Events (participants affected / at risk) | 0/261 | 0/250

LIMITATIONS AND CAVEATS:
Samples were recruited from community probation and residential probation substance abuse treatment centers. Attrition in both samples due to absconding (higher in community sample) and loss of contact with the participants in community sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT02777086/Prot_SAP_000.pdf